CLINICAL TRIAL: NCT03164057
Title: A Phase II Trial of Epigenetic Priming in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Trial of Epigenetic Priming in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML16; NCI-2017-00928 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: DNA methyltransferase inhibitors; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Decitabine; Cytarabine; Daunorubicin; Etoposide; etoposide phosphate; Methotrexate; Idarubicin; fludarabine; fludarabine phosphate; Mitoxantrone; asparaginase erwinia chrysanthemi recombinant; Sorafenib; Granulocyte Colony-Stimulating Factor; Filgrastim; Dexrazoxane; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- AZA+ADE | AZA+FLAG+Ida | AE | MA (Experimental): Part 1 Tolerability with AZA - Low Risk
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and then receive low-risk intensifications I & II without azacitidine.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide,dexrazoxane, fludarabine, idarubicin, G-CSF, mitoxantrone., ITMHA.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: G-CSF; Drug: Dexrazoxane
- DAC+ADE | DAC+FLAG+Ida | AE | MA (Experimental): Part 1 Tolerability with DAC - Low Risk
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and then receive low-risk Intensifications I & II without decitabine.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: G-CSF; Drug: Dexrazoxane
- AZA+ADE | AZA+FLAG+Ida+Sor | AZA+AE+Sor | AZA+MA+Sor (Experimental): Part 2 Dose Expansion with AZA - Low Risk
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and low- risk Intensifications I & II. Sorafenib will be given to patients with FLT3-ITD. For these patients, AZA will be limited to the first two courses of Induction chemotherapy. They will not receive AZA with Intensification therapy.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, ITMHA.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane
- DAC+ADE | DAC+FLAG+Ida+Sor | DAC+AE+Sor|DAC+MA+Sor (Experimental): Part 2 Dose Expansion with DAC - Low Risk
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and low-risk Intensifications I & II. Sorafenib will be given to patients with FLT3-ITD. For these patients, DAC will be limited to the first two courses of Induction chemotherapy. They will not receive DAC with Intensification therapy.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane
- AZA+ADE | AZA+FLAG+Ida | AE | MA | Asp+AraC (Experimental): Part 1 Tolerability with AZA - Intermediate Risk
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and then receive intermediate risk Intensifications I, II & III without azacitidine.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, erwinia asparaginase, ITMHA,
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: G-CSF; Drug: Dexrazoxane
- DAC+ADE | DAC+FLAG+Ida | AE | MA | Asp+AraC (Experimental): Part 1 Tolerability with DAC - Intermediate Risk
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and then receive intermediate-risk Intensifications I, II & III without decitabine.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, erwinia asparaginase, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: G-CSF; Drug: Dexrazoxane
- AZA| +ADE | +FLAG+Ida+Sor| +AE+Sor| +MA+Sor| +Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with AZA - Intermediate-Risk
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and intermediate-risk Intensification I, II, and III. Sorafenib will be given to patients with FLT3-ITD. For these patients, AZA will be limited to the first two courses of Induction chemotherapy. They will not receive AZA with Intensification therapy.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, asparaginase erwinia chrysanthemi (recombinant)-rywn, ITMHA.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Drug: Asparaginase Erwinia Chrysanthemi, Recombinant-Rywn
- DAC|+ADE | +FLAG+Ida+Sor | +AE+Sor | +MA+Sor | +Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with DAC - Intermediate-Risk
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and intermediate-risk Intensifications I, II and III. Sorafenib will be given to patients with FLT3-ITD. For these patients, DAC will be limited to the first two courses of Induction chemotherapy. They will not receive DAC with Intensification therapy.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, asparaginase erwinia chrysanthemi (recombinant)-rywn, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Drug: Asparaginase Erwinia Chrysanthemi, Recombinant-Rywn
- AZA+ADE | AZA+FLAG-Ida+Sor | AE | MA+Sor | Asp+AraC+Sor (Experimental): Part 1 Tolerability with AZA - High Risk (no donor)
  Patients are randomized to receive 5 days of single agent azacitidine as part of Induction I & II and high-risk intensifications I, II & III without azacitidine. Sorafenib is limited to patients with FLT3-ITD+/NUP98-NSD1+ or FLT3-ITD+/WT1mut somatic mutations.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, ITMHA.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane
- DAC+ADE | DAC+FLAG+Ida+Sor | AE | MA+Sor | Asp+AraC+Sor (Experimental): Part 1 Tolerability with DAC - High Risk (no donor)
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and then receive high-risk Intensifications I, II & III without decitabine. Sorafenib is limited to patients with FLT3-ITD+/NUP98-NSD1+ or FLT3-ITD+/WT1mut somatic mutations.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane
- AZA | + ADE | +FLAG+Ida+Sor| +AE+Sor | +MA+Sor | +Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with AZA - High Risk (no donor)
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and high-risk Intensifications I, II and III. Sorafenib will be given to patients with FLT3-ITD. For these patients, AZA will be limited to the first two courses of Induction chemotherapy. They will not receive AZA with Intensification therapy.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, asparaginase erwinia chrysanthemi (recombinant)-rywn, ITMHA.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Drug: Asparaginase Erwinia Chrysanthemi, Recombinant-Rywn
- DAC |+ADE |+FLAG+Ida+Sor |+AE+Sor|+MA+Sor|+Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with DAC - High Risk (no donor)
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and high-risk Intensifications I, II and III. Sorafenib will be given to patients with FLT3-ITD. For these patients, DAC will be limited to the first two courses of Induction chemotherapy. They will not receive DAC with Intensification therapy.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, sorafenib, mitoxantrone, erwinia asparaginase, asparaginase erwinia chrysanthemi (recombinant)-rywn, ITMHA.
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Drug: Asparaginase Erwinia Chrysanthemi, Recombinant-Rywn
- AZA+ADE | AZA+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor (Experimental): Part 1 Tolerability with AZA- High Risk (with donor)
  Patients are randomized to receive 5 days of single agent azacitidine as part of Induction I Induction II and high-risk Intensifications I or high risk intensification III without azacitidine. Patients will proceed to stem cell transplant. Sorafenib is limited to patients with FLT3-ITD+/NUP98-NSD1+ or FLT3-ITD+/WT1mut somatic mutations.
  Interventions: azacitidine cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, sorafenib, ITMHA, erwinia asparaginase, stem cell transplant.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Biological: Stem Cell Transplant
- DAC+ADE | DAC+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor (Experimental): Part 1 Tolerability with DAC - High Risk (with donor)
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and then receive high-risk Intensifications I or high risk intensification III without decitabine. Patients will proceed to stem cell transplant. Sorafenib is limited to patients with FLT3-ITD+/NUP98-NSD1+ or FLT3-ITD+/WT1mut somatic mutations.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, sorafenib, ITMHA, erwinia asparaginase, stem cell transplant
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Biological: Stem Cell Transplant
- DAC |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with DAC - High Risk (with donor)
  Patients are randomized to receive 5 days of single agent decitabine as part of Inductions I & II and high-risk Intensifications I or high risk intensification III. Patients will proceed to stem cell transplant. Sorafenib will be given to patients with FLT3-ITD. For these patients, DAC will be limited to the first two courses of Induction chemotherapy. They will not receive DAC with Intensification therapy.
  Interventions: decitabine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G- CSF, mitoxantrone, sorafenib, ITMHA, erwinia asparaginase, stem cell transplant
  Interventions: Drug: Decitabine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Biological: Stem Cell Transplant
- AZA |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor (Experimental): Part 2 Dose Expansion with AZA - High Risk (with donor)
  Patients are randomized to receive 5 days of single agent azacitidine as part of Inductions I & II and high-risk Intensification I or high risk intensification III. Patients will proceed to stem cell transplant. Sorafenib will be given to patients with FLT3-ITD. For these patients, AZA will be limited to the first two courses of Induction chemotherapy. They will not receive AZA with Intensification therapy.
  Interventions: azacitidine, cytarabine, daunorubicin, etoposide, dexrazoxane, fludarabine, idarubicin, G-CSF, mitoxantrone, sorafenib, ITMHA, erwinia asparaginase, stem cell transplant.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Combination Product: ITMHA; Drug: Idarubicin; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Erwinia asparaginase; Drug: Sorafenib; Drug: G-CSF; Drug: Dexrazoxane; Biological: Stem Cell Transplant

INTERVENTIONS:
Drug: Azacitidine — Azacitidine solution is administered intravenously (IV) over a period of 10-40 minutes.
  Other Names: Vidaza®
  Arms: AZA | + ADE | +FLAG+Ida+Sor| +AE+Sor | +MA+Sor | +Asp+AraC+Sor; AZA |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; AZA+ADE | AZA+FLAG+Ida | AE | MA; AZA+ADE | AZA+FLAG+Ida | AE | MA | Asp+AraC; AZA+ADE | AZA+FLAG+Ida+Sor | AZA+AE+Sor | AZA+MA+Sor; AZA+ADE | AZA+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; AZA+ADE | AZA+FLAG-Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; AZA| +ADE | +FLAG+Ida+Sor| +AE+Sor| +MA+Sor| +Asp+AraC+Sor
Drug: Decitabine — Administered intravenously (IV) over approximately one hour.
  Other Names: Dacogen®
  Arms: DAC |+ADE |+FLAG+Ida+Sor |+AE+Sor|+MA+Sor|+Asp+AraC+Sor; DAC |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida | AE | MA; DAC+ADE | DAC+FLAG+Ida | AE | MA | Asp+AraC; DAC+ADE | DAC+FLAG+Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | DAC+AE+Sor|DAC+MA+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; DAC|+ADE | +FLAG+Ida+Sor | +AE+Sor | +MA+Sor | +Asp+AraC+Sor
Drug: Cytarabine — Given IV or intrathecally (IT).
  Other Names: Ara-C; Cytosar®
Drug: Daunorubicin — Given IV.
  Other Names: Daunomycin; Cerubidine®
Drug: Etoposide — Given IV.
  Other Names: Vepesid®; VP-16; Etoposide Phosphate; Etopophos®
Combination Product: ITMHA — Given IT.
  Other Names: Intrathecal Triples; Methotrexate/Hydrocortisone/Cytarabine
Drug: Idarubicin — Given IV.
  Other Names: Idamycin PFS®
Drug: Fludarabine — Given IV over approximately 30 minutes.
  Other Names: Fludara®
Drug: Mitoxantrone — Given IV.
  Other Names: Novantrone®
Drug: Erwinia asparaginase — Given IV or intramuscularly (IM).
  Other Names: Asparaginase Erwinia chrysanthemi; Erwinaze®; Crisantaspase®
  Arms: AZA | + ADE | +FLAG+Ida+Sor| +AE+Sor | +MA+Sor | +Asp+AraC+Sor; AZA |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; AZA+ADE | AZA+FLAG+Ida | AE | MA | Asp+AraC; AZA+ADE | AZA+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; AZA+ADE | AZA+FLAG-Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; AZA| +ADE | +FLAG+Ida+Sor| +AE+Sor| +MA+Sor| +Asp+AraC+Sor; DAC |+ADE |+FLAG+Ida+Sor |+AE+Sor|+MA+Sor|+Asp+AraC+Sor; DAC |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida | AE | MA | Asp+AraC; DAC+ADE | DAC+FLAG+Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; DAC|+ADE | +FLAG+Ida+Sor | +AE+Sor | +MA+Sor | +Asp+AraC+Sor
Drug: Sorafenib — Given PO.
  Other Names: Nexavar®
  Arms: AZA | + ADE | +FLAG+Ida+Sor| +AE+Sor | +MA+Sor | +Asp+AraC+Sor; AZA |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; AZA+ADE | AZA+FLAG+Ida+Sor | AZA+AE+Sor | AZA+MA+Sor; AZA+ADE | AZA+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; AZA+ADE | AZA+FLAG-Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; AZA| +ADE | +FLAG+Ida+Sor| +AE+Sor| +MA+Sor| +Asp+AraC+Sor; DAC |+ADE |+FLAG+Ida+Sor |+AE+Sor|+MA+Sor|+Asp+AraC+Sor; DAC |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | AE | MA+Sor | Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | DAC+AE+Sor|DAC+MA+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; DAC|+ADE | +FLAG+Ida+Sor | +AE+Sor | +MA+Sor | +Asp+AraC+Sor
Drug: G-CSF — Given IV.
  Other Names: Neupogen; Filgrastim
Drug: Dexrazoxane — Given IV immediately before idarubicin administration.
  Other Names: Zinecard®
Biological: Stem Cell Transplant — The transplant protocol will depend on the patient's donor and transplant physician's preference.
  Other Names: SCT
  Arms: AZA |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; AZA+ADE | AZA+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor; DAC |+ADE|+FLAG+Ida+Sor|+MA+Sor|+Asp+AraC+Sor; DAC+ADE | DAC+FLAG+Ida+Sor | MA+Sor | Asp+AraC+Sor
Drug: Asparaginase Erwinia Chrysanthemi, Recombinant-Rywn — May be used in the event of an Erwinia asparaginase shortage. Given intramuscularly (IM).
  Other Names: Rylaze™; Recombinant Erwinia
  Arms: AZA | + ADE | +FLAG+Ida+Sor| +AE+Sor | +MA+Sor | +Asp+AraC+Sor; AZA| +ADE | +FLAG+Ida+Sor| +AE+Sor| +MA+Sor| +Asp+AraC+Sor; DAC |+ADE |+FLAG+Ida+Sor |+AE+Sor|+MA+Sor|+Asp+AraC+Sor; DAC|+ADE | +FLAG+Ida+Sor | +AE+Sor | +MA+Sor | +Asp+AraC+Sor

SUMMARY:
The overall aim of this study is to determine if epigenetic priming with a DNA methyltransferase inhibitor (DMTi) prior to chemotherapy blocks is tolerable and carries evidence of a clinical efficacy signal as determined by minimal residual disease (MRD), event-free survival (EFS), and overall survival (OS). Tolerability for each of the agents, as well as total reduction in DNA methylation and outcome assessments will be done to simultaneously obtain preliminary biological and clinical data for each DMTi in parallel.

PRIMARY OBJECTIVES:

* Evaluate the tolerability of five days of epigenetic priming with azacitidine and decitabine as a single agent DMTi prior to standard AML chemotherapy blocks.
* Evaluate the change in genome-wide methylation burden induced by five days of epigenetic priming and the association of post-priming genome-wide methylation burden with event-free survival among pediatric AML patients.

SECONDARY OBJECTIVES

* Describe minimal residual disease levels following Induction I chemotherapy in patients that receive DMTi.
* Estimate the event-free survival and overall survival of patients receiving a DMTi prior to chemotherapy courses.

DETAILED DESCRIPTION:
To determine tolerability, priming with DMTi (azacitidine or decitabine) will be limited to Induction I and II during Part 1 of the study. If DMTi treatment is tolerated during Part 1, the investigators will go on to an Expansion Phase (Part 2) that includes DMTi priming prior to all chemotherapy blocks.

Treatment will consist of 5 blocks of conventional chemotherapy: Induction I, Induction II, Intensification I, Intensification II, and Intensification III over approximately 5 months.

RANDOMIZATION: Patients will be randomized to receive one of two DMTi (azacitidine or decitabine) for 5 days prior to Induction I. Intrathecal (ITHMA) treatments will be given right before treatment on this study or on Day 1 of Induction I treatment. Leucovorin will be given 24-30 hours following ITHMA.

INDUCTION I CHEMOTHERAPY: Patients receive cytarabine, daunorubicin, and etoposide.

INDUCTION II CHEMOTHERAPY; Patients receive their assigned DMTi for 5 days followed by fludarabine, cytarabine, G-CSF, and idarubicin.

Patients are then evaluated and assigned to either the low-risk arm, intermediate-risk arm, or the high-risk arm for Intensification therapy.

Patients with ≥ 5% blasts following Induction II will be considered refractory and will go off therapy. The rare high risk patient with an MRD < 0.1% following Induction I may proceed directly to stem cell transplant (SCT) after Induction II - if a suitable donor is available and the transplant can be performed without delay. MDS patients may proceed to SCT once they have achieved MRD <0.1% irrespective of the number of chemotherapy courses received.

INTENSIFICATION I CHEMOTHERAPY - LOW-RISK AML, INTERMEDIATE-RISK AML, and HIGH-RISK AML with no donor: Patients receive cytarabine and etoposide. After administration of 5 days of a DMTi prior to Inductions I and II satisfies a tolerability determination criterion, patients will also receive their randomly assigned DMTi for five days prior to cytarabine and etoposide.

INTENSIFICATION II CHEMOTHERAPY - LOW RISK AML, INTERMEDIATE-RISK AML, and HIGH-RISK AML with no donor: Patients receive mitoxantrone and cytarabine. After administration of 5 days of a DMTi prior to Inductions I and II satisfies a tolerability determination criterion, patients will also receive their randomly assigned DMTi for five days prior to mitoxantrone and cytarabine.

INTENSIFICATION I CHEMOTHERAPY - HIGH-RISK AML with a donor: Patients receive mitoxantrone and cytarabine followed by stem cell transplant (SCT). Treatment related AML patients and patients with treatment related MDS who have a donor but are not able to receive a SCT without delay will proceed to HR Intensification III and receive erwinia asparaginase and cytarabine. After administration of 5 days of a DMTi prior to earlier courses satisfies a tolerability criterion, patients will also receive their randomly assigned DMTi for five days prior to mitoxantrone and cytarabine or erwinia asparaginase and cytarabine.

Treatment related AML patients and treatment related MDS patients that are not able to receive a SCT should go off treatment following Intensification II.

INTENSIFICATION III CHEMOTHERAPY - INTERMEDIATE-RISK AML and HIGH-RISK AML with no donor: Patients receive erwinia asparaginase and cytarabine. After administration of 5 days of a DMTi prior to earlier courses satisfies a tolerability criterion, patients will also receive their randomly assigned DMTi for five days prior to erwinia asparaginase and cytarabine.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnostic criteria: Patients must have one of the following diagnoses:

  * Acute myeloid leukemia fulfilling the criteria of the WHO Classification (see Appendix I), or
  * >5% but < 20% marrow myeloblasts and evidence of a clonal de novo AML genetic abnormality [e.g., t(8;21), inv(16), t(9;11)], or
  * Myeloid sarcoma (also referred to as extramedullary myeloid tumor, granulocytic sarcoma, or chloroma), with or without evidence of a leukemia process in the bone marrow or peripheral blood, with confirmation of myeloid differentiation, or
  * High grade myelodysplastic syndrome (MDS) with greater than 5% blasts, or
  * Patients with treatment related myeloid neoplasms including AML and MDS, provided their cumulative anthracycline dose has not exceeded 230 mg/m2 doxorubicin equivalents.
* Other criteria - Patients must meet all the following criteria:

  * Age > 28 days and < 22 years at time of study entry inclusive, and
  * No prior therapy for this malignancy except for one dose of intrathecal therapy and the use of hydroxyurea or low-dose cytarabine (100-200 mg/m2 per day for one week or less for hyperleukocytosis), and
  * Written informed consent according to institutional guidelines, and
  * Female patients of childbearing potential must have a negative pregnancy test within 2 weeks prior to enrollment, and
  * Male and female participants of reproductive potential must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

EXCLUSION CRITERIA:

* Down syndrome
* Acute promyelocytic leukemia (APL)
* BCR-ABL1 chronic myeloid leukemia in blast crisis (CML-BC)
* Juvenile myelomonocytic leukemia (JMML)
* Fanconi anemia (FA)
* Kostmann syndrome
* Shwachman syndrome
* Other bone marrow failure syndromes or low grade (<5% bone marrow blasts) MDS.
* Use of concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy for this malignancy within 2 weeks before study entry with the exception of IT therapy, hydroxyurea, or low-dose cytarabine as specified in the protocol document. The patient must have recovered from all acute toxicities from any previous therapy.
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Prior chemotherapy, with the exception of hydroxyurea or low-dose cytarabine as specified in the protocol document. The patient must have recovered from all acute toxicities from any previous therapy.
* Patients with treatment related myeloid neoplasms with cumulative anthracyclines greater than 230 mg/m2 doxorubicin equivalents.

Ages: 29 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 206 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of evaluable patients who tolerate five days of single agent DMTi before a standard chemotherapy combination | From enrollment to completion of chemotherapy (up to 8 months after start of therapy)
  Patients will be monitored for grade 4-5 non-hematologic toxic events during these two courses of chemotherapy. Tolerating a course is defined as completing the course without experiencing death or a grade 4 non-hematologic toxicity.
Change in genome-wide methylation burden of leukemia cells from diagnosis to after five days of single agent DMTi | From diagnosis to completion of five days of single agent DMTi (up to 2 weeks after start of therapy)
  Leukemic cells will be collected from patients at diagnosis and after five days of single agent DMTi. Each sample of leukemic cells will be profiled with a methylation microarray. For each leukemic sample, genome-wide methylation burden (GWMB) will be computed as the sum of methylation values across all markers. For each patient, the change in GWMB will be computed as the day 5 GWMB minus the diagnostic GWMB.
Cox model hazard ratio for association of event-free survival with genome-wide methylation burden | From diagnosis to the first of the following events: death, relapse, resistant disease, second malignancy, or last follow-up (up to 3 years after completion of therapy)
  Patients will be monitored for the events of interest from enrollment for at least three years. EFS will be defined as the time elapsed from enrollment to the first of the following events: death, relapse, resistant disease, or second malignancy. EFS times for subjects who have not experienced these events at the time of analysis will be censored at date of last follow-up. A Cox regression model will be used to evaluate the association of EFS with genome-wide methylation burden observed after completion of five days of single agent decitabine or azacitidine as randomly assigned.

SECONDARY OUTCOMES:
Proportion of MRD-evaluable subjects with detectable minimal residual disease after receiving five days of a single agent DMTi followed by araC+daunorubicin+etoposide. | MRD will be measured after completion of DMTi+araC+daunorubicin+etoposide (up to 6 weeks after the start of therapy)
  Flow cytometry will be used to measure minimal residual disease at diagnosis and after completion of the first course of chemotherapy.
Kaplan-Meier estimate of event-free survival | From diagnosis to the first of the following events: death, relapse, resistant disease, second malignancy, or last follow-up (up to 3 years after completion of therapy)
  Patients will be monitored for the events of interest from enrollment for at least three years. EFS will be defined as the time elapsed from enrollment to the first of the following events: death, relapse, resistant disease, or second malignancy. EFS times for subjects who have not experienced these events at the time of analysis will be censored at date of last follow-up.
Kaplan-Meier estimate of overall survival | From diagnosis to the first of the following events: death or last follow-up (up to 3 years after completion of therapy)
  Patients will be monitored for death from enrollment for at least three years. Overall survival will be defined as the time elapsed from enrollment to death. OS times for subjects who are living at the time of analysis will be censored at date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Raul C. Ribiero, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (10):
- United States (10):
  - Children's Hospital of Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital and Health Center, San Diego, California
  - University of Chicago Children's Hospital (Comer), Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols